CLINICAL TRIAL: NCT04385693
Title: Intentional Pulpotomy to Preserve Vital Primary Molars With Challenging Restorability: a Feasibility Study
Brief Title: Intentional Pulpotomy to Preserve Hopeless Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: NuSmile, Ltd and Avalon Biomed (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202000068; OCR34882 (Other: UF OnCore)
Record Dates: First submitted 2020-05-01; First posted 2020-05-13 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Pulpitis; Dental Pulp Diseases; Tooth Diseases
MeSH Terms: conditions — Pulpitis; Dental Pulp Diseases; Tooth Diseases | interventions — Pulpotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): Group A: The patient will benefit from an experimental treatment: a Pulpotomy. The pulpotomy aims at removing the coronal part of the pulp (the pulp present in the pulp chamber) and filling the pulp chamber with a bioactive material.
  Interventions: Procedure: Pulpotomy
- Control Group (Active Comparator): Group B: Extracted teeth will serve as controls, and information regarding the need or not of space maintenance, and the impact on the occlusion and eruption of the succedaneous permanent tooth will be noted.
  Interventions: Procedure: Extraction and placement of space maintainer

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy using bioactive bioceramic cement of 1.5 mm layer of a newly FDA approved calcium-based silicate cement (Nusmile NeoPutty) will be placed on the pulp chamber floor and canals' orifices for pulp and root therapy. Pulpotomy is a procedure in which the coronal pulp is amputated, and the remaining radicular pulp tissue is treated with a medicament to preserve the pulp's health.This technique involves administration of local analgesia, Isolation of the tooth with rubber dam, complete caries removal and then access to the pulp chamber using drills.
  Arms: Pulpotomy
Procedure: Extraction and placement of space maintainer — If during the pulpotomy procedure, hemostasis is not obtainable, or signs of advanced pulp degeneration such as dark and limited or no bleeding from canals, the pulp will be diagnosed as chronically inflamed or necrotic, and tooth will be extracted. As part of the standard of care after extractions of primary molars, space maintenance will be assessed, and a space maintainer fabricated if indicated. Extracted teeth will serve as controls, and information regarding the need or not of space maintenance.
  Arms: Control Group

SUMMARY:
When proximal carious lesions of primary molars are located in close proximity to the cementum enamel junction (CEJ), marginal seal is challenging and extraction is recommended. Pulpotomy is indicated for vital primary teeth to preserve them in function. The goal of this study is to monitor the long-term effect of intentional bioactive cement pulpotomies and crown coverage performed on vital and asymptomatic carious primary molars with gingival margins close to or at the CEJ

ELIGIBILITY:
Inclusion Criteria:

* Selected patients will have one or more primary molar teeth diagnosed clinically with large proximal carious lesions with the gingival extension of the cavity at or below the cemento-enamel junction. The tooth should be asymptomatic and must have no signs of swelling, fistula, abnormal mobility and sensitivity to percussion (ruling out food impaction), and adequate space for placement of a stainless steel crown restoration. The pre-operative periapical radiograph, taken as part of the new patient/recall routine visit, should reveal a lesion in close approximation to the pulp, but having at least 1-2 mm of sound dentin separating the deepest portion of the lesion and the pulp. In addition, no evidence of furcation and periapical pathology, internal or external root resorption and presence of half to two-thirds of root length remaining.

Exclusion Criteria:

* Uncooperative patients
* Teeth with positive history of pain, abnormal mobility, signs of pulp necrosis such as presence of swelling or fistula, and significant space loss due to caries not allowing placement of a stainless steel crown restoration
* Radiographically, signs of furcation and periapical pathology, internal and external resorption, less than half to 2/3 of root length remaining
* Selected patients will be treated by pediatric dental residents in the regular dental clinic setting with or without nitrous oxide inhalation, as part of the standard of care
* Prior to the beginning of the study, all operators will be calibrated by the principal investigator on identifying the teeth in question, as well as on the restorative technique
* Selected patients may have one or more qualified teeth

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Radiographic examination for each recall visit | up to 1 year
  Evaluation of asymptomatic tooth in the mouth for presence of infection (bite -wing/periapical radiograph(s)

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Guelmann, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No